CLINICAL TRIAL: NCT01109524
Title: Cisplatin and Vinorelbine in Combination With Cetuximab as First Line Treatment for Patients With Advanced/Metastatic Non-Small Cell Lung Cancer (NSCLC): a Single Arm Multicenter Safety Phase 2 Study
Brief Title: Safety Study of Cetuximab in Combination With Cisplatin and Vinorelbine to Treat Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA225-346
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Lung Neoplasms; Carcinoma; Cancer of the Lung; Non-Small-Cell Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms; Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Cisplatin; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab + Cisplatin + Vinorelbine (Experimental)
  Interventions: Drug: Cetuximab; Drug: Cisplatin; Drug: Vinorelbine

INTERVENTIONS:
Drug: Cetuximab — Vial, Intravenous, 400mg/m², week 1, then 250mg/m², Weekly, Until Progressive Disease (PD)/ Toxicity/Pt-PI Decision
  Other Names: Erbitux; BMS-564717
Drug: Cisplatin — Vial, Intravenous, 80mg/m², Day 1 of each 21 day cycle, Maximum 6 cycles
  Other Names: Platinol
Drug: Vinorelbine — Vial, Intravenous, 25 mg/m², Day 1 and 8 of each 21 day cycle, Maximum 6 cycles
  Other Names: Navelbine

SUMMARY:
The purpose of the study is to determine if U.S. manufactured Cetuximab can be safely used for the treatment of Non-Small Cell Lung Cancer in combination with Cisplatin and Vinorelbine.

ELIGIBILITY:
Inclusion Criteria:

* Non-Small Cell Lung Cancer (NSCLC), Stage IV (per the American Joint Committee on Cancer (AJCC) Staging Manual, Seventh Edition) or recurrent disease following surgery and/or radiation therapy
* Evaluable or measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2

Exclusion Criteria:

* Uncontrolled Central Nervous System (CNS) metastasis.
* Previous exposure to monoclonal antibodies, signal transduction inhibitors or Epidermal growth factor receptor (EGFR) targeting therapy
* Concurrent malignancy
* Prior chemotherapy for NSCLC
* Pre-existing ascites grade ≥ 2 or pericardial effusion grade ≥ 2
* Superior vena cava syndrome contra-indicating hydration
* White Blood Cells (WBC) < 3,000/mm³
* Absolute neutrophile count (ANC) < 1,500/mm³
* Platelet < 100,000/mm³
* Hemoglobin (Hgb) < 9.0 g/dL
* Total bilirubin > 1.5 x Upper limit of normal (ULN).
* Aspartate aminotransferase (AST) or Alanine-aminotransferase (ALT) > 5.0 x ULN.
* Serum creatinine >1.25 x ULN and calculated creatinine clearance <60mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (22):
- United States (13):
  - Donald W. Hill M.D., P.C., Casa Grande, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Cancer Care Institute, Los Angeles, California
  - Northern California Hematology & Oncology, Oakland, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Broward Oncology Associates, P.A., Fort Lauderdale, Florida
  - Elite Research Institute, Miami, Florida
  - Edward H. Kaplan, MD & Associates, Skokie, Illinois
  - Fairview Southdale Medical Oncology Clinic, Edina, Minnesota
  - Mid Dakota Clinic, Pc, Bismarck, North Dakota
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University Medical Center, Lubbock, Texas
  - Columbia Basin Hematology and Oncology, Kennewick, Washington
- Canada (7):
  - The Moncton Hospital, Moncton, New Brunswick
  - Local Institution, Grand Falls-Windsor, Newfoundland and Labrador
  - Sudbury Regional Hospital, Greater Sudbury, Ontario
  - The Credit Valley Hospital, Mississauga, Ontario
  - Thunder Bay Regional Health Sciences Centre (Regional Cancer Care), Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Centre de sante et de services sociaux de Rimouski-Neigette, Rimouski, Quebec
- Puerto Rico (2):
  - Ponce School of Medicine (Caimed Center), Ponce
  - Fundacion de Investigacion de Diego, San Juan

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant, first visit: 1 July 2010; Last participant, last visit: 7 September 2012. Participants were chemotherapy-naive with Stage IV histologically or cytologically documented non-small cell lung cancer (NSCLC). Participants treated until: progressive disease (PD)/ toxicity/patient-investigator decision.
Pre-assignment Details: 72 participants were enrolled and 60 were treated with study drug. 12 not treated: 10 participants no longer met study criteria and 2 participants withdrew consent before entering the treatment phase.
Groups:
- Cetuximab + Cisplatin/Vinorelbine: Intravenous (IV) cetuximab, 400mg per meter^2 (m^2), Week 1, then 250mg/m^2 weekly, until progressive disease (PD) or toxicity or participant-principal investigator (PPI)decision stopped treatment. One hour of observation required after each infusion. Cisplatin administered as IV solution at initial dose of 80mg/m^2 on the first day of each 21 day treatment cycle. Vinorelbine administered as IV solution at initial dose of 25 mg/m^2 on Day 1 and Day 8 of each 21 day treatment cycle. One cycle was defined as a 21-day treatment period, unless chemotherapy administration was delayed (cycle duration was longer). All study drugs discontinued if participants experienced PD. If unacceptable toxicities to any study drug occurred, any drug could be modified (reduced, delayed, omitted, or discontinued) independently of the other drugs If no PD, cetuximab could be given as monotherapy after completion of the 6 treatment cycles or after early discontinuation of cis/vin due to intolerance.
Period: Overall Study
Arm/Group | Cetuximab + Cisplatin/Vinorelbine
Started | 60
Completed | 3
Not Completed | 57
Not completed — Disease Progression | 29
Not completed — Study Drug toxicity | 6
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 2
Not completed — Maximum clinical benefit | 3
Not completed — Death | 2
Not completed — No longer meets criteria | 2
Not completed — Participant requested to end treatment | 4
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Population: All treated participants.
Groups:
- Cetuximab + Cisplatin/Vinorelbine: Intravenous (IV) cetuximab, 400mg per meter^2 (m^2), Week 1, then 250mg/m^2 weekly, until progressive disease (PD) or toxicity or participant-principal investigator (PPI) decision stopped treatment. One hour of observation required after each infusion. Cisplatin administered as IV solution at initial dose of 80mg/m^2 on the first day of each 21 day treatment cycle. Vinorelbine administered as IV solution at initial dose of 25 mg/m^2 on Day 1 and Day 8 of each 21 day treatment cycle. One cycle was defined as a 21-day treatment period, unless chemotherapy administration was delayed (cycle duration was longer). All study drugs discontinued if participants experienced PD. If unacceptable toxicities to any study drug occurred, any drug could be modified (reduced, delayed, omitted, or discontinued) independently of the other drugs If no PD, cetuximab could be given as monotherapy after completion of the 6 treatment cycles or after early discontinuation of cis/vin due to intolerance.
Arm/Group | Cetuximab + Cisplatin/Vinorelbine
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 23
  Puerto Rico | 7
  Canada | 30
ECOG PS at baseline [Number; unit: Participants] — ECOG PS = Eastern Cooperative Oncology Group Performance Status. Baseline is defined as values obtained during the screening period, prior to treatment with study drug. Inclusion criteria included those participants with values of 0, 1 or 2. ECOG=performance questionnaire with a scale of 6 units (0 to 5) with the higher numbers reflecting a worse outcome: 0=fully active, carry on performance without restriction; 1=restricted in physically strenuous activity but ambulatory, 2= ambulatory and capable of self care; 3=capable of limited self care, confined to bed; 4=completely disabled; 5=dead.
  Participants
    0 | 17
    1 | 38
    2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths, and AEs Leading to Discontinuation of at Least One Study Drug, - Treated Population
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=medical event that results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. MedDRA version 14.0. Severity of AEs were graded according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 3.0: Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Life-threatening or disabling, Gr 5=Death. Day 1 (start of study drug) to 30 days after last dose of any treatment therapy, including cetuximab monotherapy.
Time Frame: Day 1 up to 30 days after last dose
Population: Treated population: all participants who received at least one dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Cetuximab + Cisplatin/Vinorelbine
Number analyzed (Participants) | 60
participants
  Deaths due to disease progression | 3
  Deaths due to Other Causes | 2
  SAE (any grade) | 38
  AE (any grade) | 59
  AE Grade 3 or 4 | 46
  AE that led to Discontinuation of study drug | 21

2. Primary Outcome: Number of Participants With Grades 3 and 4 Treatment-emergent Adverse Events (AEs) of Special Interest - Treated Population
Description: Special interest AEs: acneform rash, infusion reaction, cardiac adverse event, febrile neutropenia, infection (includes all terms except sepsis), sepsis, interstitial lung disease, renal failure, and thromboembolic events. Except for interstitial lung disease, these were composite terms combining several preferred/other level MedDRA terms (MedDRA version 14.0). Except for Grade (GR)3 and 4 infusion reactions, AE severity were graded per the NCI-CTC, version 3.0: Gr 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Life-threatening or disabling, Gr 5=Death. Severity of Gr 3 - 4 infusion reactions were: Gr 3=symptomatic bronchospasm, requiring parenteral medication(s), with or without urticaria; allergy-related edema/angioedema; Gr 4=a life-threatening event characterized by the same symptomatology as a Gr 3, complicated by symptomatic hypotension or oxygen saturation 70% or less. Day 1 (start of study drug) to 30 days after last dose of any treatment therapy, including cetuximab monotherapy.
Time Frame: Day 1 to 30 days after last dose
Population: Treated population: all participants who received at least one dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Cetuximab + Cisplatin/Vinorelbine
Number analyzed (Participants) | 60
participants
  Grade 3-4 acneform rash | 5
  Grade 3-4 infusion reaction | 2
  Cardiac events Grade 3-4 | 3
  Infection Grade 3-4 | 9
  Sepsis Grade 3-4 | 0
  Renal failure Grade 3-4 | 3
  Thromboembolic events Grade 3-4 | 11
  Interstitial lung disease Grade 3-4 | 0
  Febrile neutropenia Grade 3-4 | 6

3. Primary Outcome: Number of Participants With Liver Function Serum Chemistry Laboratory Abnormalities - Treated Population
Description: ULN=Upper limit of normal among all laboratory ranges. ALT=alanine transaminase; AST=aspartate aminotransferase; ALP=alkaline phosphatase. CTC grade criteria: ALT Grade 1:>ULN 2.5*ULN; Grade 2: >2.5 - 5.0*ULN; Grade 3: >5.0 - 20.0*ULN; Grade 4: >20.0*ULN. AST Grade 1: >ULN - 2.5*ULN; Grade 2: >2.5 - 5.0*ULN; Grade 3: >5.0 - 20.0*ULN; Grade 4: >20.0*ULN. Total bilirubin Grade 1: >ULN - 1.5*ULN; Grade 2: >1.5 - 3.0*ULN; Grade 3: >3.0 - 10.0*ULN; Grade 4: >10.0*ULN. Albumin (low) Grade 1:<LLN - 3 grams per deciliter (g/dL)to <LLN - 3 g/dL; Grade 2: <3 - 2 g/dL to < 3.0 - 2.0 g/dL; Grade 3: < 2 g/dL to <2 g/L. Day 1 (start of study drug) to 30 days after last dose of any treatment therapy, including cetuximab monotherapy.
Time Frame: Day 1 up to 30 days after last dose
Population: Number (N) of participants with laboratory data available and who could be analyzed for total bilirubin was 49. All other liver function laboratories N=57. Treated population: all participants who received at least one dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Cetuximab + Cisplatin/Vinorelbine
Number analyzed (Participants) | 57
participants
  Albumin (low) Grade 1 - 4 | 37
  Albumin (low) Grade 3 or 4 | 0
  Total bilirubin (high) Grade 1 - 4 (N=49) | 3
  Total bilirubin (high) Grade 3 or 4 (N=49) | 0
  ALT (high) Grade 1 - 4 | 31
  ALT (high) Grade 3 or 4 | 0
  ALP (high) Grade 1 - 4 | 26
  ALP (high) Grade 3 or 4 | 0
  AST (high) Grade 1 - 4 | 19
  AST (high) Grade 3 or 4 | 0

4. Primary Outcome: Number of Participants With Hematology Laboratory Abnormalities - Treated Population
Description: Hematology laboratories included hemoglobin, platelets, white blood cell (WBC) count, and absolute neutrophil count (ANC) and values were per CTC grading, 0, 1, 2, 3, 4. On-study laboratory tests were those performed after the start of study drug (from Day 2 of cycle 1) and up to 30 days after the last dose of study drug. WBC normal range: 4.1-12.3 x 10^3 /microliter (µL); platelets normal range: 140-450 x 10^9 /Liter (L); hemoglobin normal range 14-18 grams per deciliter (g/dL); ANC normal range: 2.03-8.36 x 10^9/μL.
Time Frame: Day 2 up to 30 days after last dose
Population: Treated population: all participants who received at least one dose of any study drug. Participants with at least one on-study laboratory measurement available were analyzed.
Measure: Number; unit: participants
Arm/Group | Cetuximab + Cisplatin/Vinorelbine
Number analyzed (Participants) | 57
participants
  Hemoglobin (low) Grade 1 - 4 | 51
  Hemoglobin (low) Grade 3 or 4 | 4
  Hemoglobin (low) Grade 4 | 0
  Platelets (low) Grade 1 - 4 | 19
  Platelets (low) Grade 3 or 4 | 1
  Platelets (low) Grade 4 | 0
  WBC (low) Grade 1 - 4 | 49
  WBC (low) Grade 3 or 4 | 28
  WBC (low) Grade 4 | 6
  ANC (low) Grade 1 - 4 | 47
  ANC (low) Grade 3 or 4 | 38
  ANC (low) Grade 4 | 24

5. Primary Outcome: Number of Participants With Renal Function Serum Chemistry Laboratory Abnormalities - Treated Population
Description: ULN=Upper limit of normal among all laboratory ranges; LLN=Lower limit of normal. CTC grade criteria: Sodium high (H) Grade (Gr) 1:>ULN - 150 millimoles per liter (mmol/L); Gr 2: >150 - 155 mmol/L; Gr 3: >155 - 160mmol/L; Gr 4: >160 mmol/L. Sodium low(L) Gr 1:<LLN - 130mmol/L; Gr 3: <130 - 120 mmol/L; Gr 4: <120 mmol/L. Potassium (H) Gr 1: >ULN - 5.5 mmol/L; Gr 2: >5.5 - 6.0 mmol/L; Gr 3: > 6.0 - 7.0 mmol/L; Gr 4: >7.0 mmol/L. Potassium (L) Gr 1: <LLN - 3.0 mmol/L; Gr 2: <LLN - 3.0 mmol/L; Gr 3: < 3.0 - 2.5 mmol/L; Gr 4: <2.5 mmol/L. Serum creatinine (H) Gr 1: >1 - 1.5*baseline (BL)to >ULN - 1.5*ULN; Gr 2: >1.5 - 3.0*BL to > 1.5 - 3.0*ULN; Gr 3: >3.0*BL to > 3.0 - 6.0*ULN; Gr 4: >6.0*ULN. Day 1 (start of study drug) to 30 days after last dose of any study drug, including monotherapy.
Time Frame: Day 1 up to 30 days after last dose
Population: Treated population: All participants who received at least one dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Cetuximab + Cisplatin/Vinorelbine
Number analyzed (Participants) | 57
participants
  Sodium (low) Grade 1 - 4 | 42
  Sodium (low) Grade 3 or 4 | 18
  Sodium (low) Grade 4 | 0
  Sodium (high) Grade 1 - 4 | 1
  Sodium (high) Grade 3 or 4 | 0
  Sodium (high) Grade 4 | 0
  Potassium (low) Grade 1 - 4 | 29
  Potassium (low) Grade 3 or 4 | 12
  Potassium (low) Grade 4 | 1
  Potassium (high) Grade 1 - 4 | 10
  Potassium (high) Grade 3 or 4 | 1
  Potassium (high) Grade 4 | 0
  Serum Creatinine (high) Grade 1 - 4 | 15
  Serum Creatinine (high) Grade 3 or 4 | 0
  Serum Creatinine (high) Grade 4 | 0

6. Primary Outcome: Number of Participants With Drug-Related Treatment-emergent AEs, Drug-Related SAEs, and Drug-Related AEs Leading to Discontinuation of at Least One Study Drug, - Treated Population
Description: Drug-related AEs and drug-related SAEs (by investigator assessment) were those with a relationship to study drug(s) reported to Sponsor as related and those of unknown relationship. AE was defined as any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE was defined as a medical event that results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. MedDRA version 14.0. Severity of AEs were graded according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 3.0: Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Life-threatening or disabling, Gr 5=Death. Day 1 (start of study drug) to 30 days after last dose of any study drug, including monotherapy.
Time Frame: Day 1 up to 30 days after last dose
Population: Treated population: All participants who received at least one dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Cetuximab + Cisplatin/Vinorelbine
Number analyzed (Participants) | 60
participants
  Drug-related SAE (any grade) | 16
  Drug-related AE (any grade) | 54
  Drug-related AE Grade 3 or 4 | 31
  Drug-related AE led to Discontinuation of drug | 11

7. Primary Outcome: Number of Participants With Grades 3 and 4 Drug-Related Treatment-emergent AEs of Special Interest - Treated Population
Description: Drug-related AEs (investigator assessment): those with relationship to study drug(s)reported as related and those of unknown relationship. Special interest AEs: acneform rash, infusion reaction, cardiac adverse event, febrile neutropenia, infection (all terms except sepsis), sepsis, interstitial lung disease, renal failure, and thromboembolic events. Except for interstitial lung disease, these were composite terms combining several MedDRA terms (MedDRA version 14.0). Except for Gr 3 and 4 infusion reactions, AE severity per NCI-CTC, version 3.0: Gr 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Life-threatening or disabling, Gr 5=Death. Gr 3 - 4 infusion reactions: Gr 3=symptomatic bronchospasm, requiring parenteral medication(s), with or without urticaria; allergy-related edema/angioedema; Gr 4=life-threatening event with same Gr 3 symptomatology, complicated by symptomatic hypotension/oxygen saturation 70% or less. Day 1=start of study drug; to 30 days after last dose of any treatment.
Time Frame: Day 1 up to 30 days after last dose
Population: Treated population: All participants who received at least one dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Cetuximab + Cisplatin/Vinorelbine
Number analyzed (Participants) | 60
participants
  drug-related acneform rash Grade 3 - 4 | 5
  drug-related infusion reaction Grade 3 - 4 | 2
  drug-related cardiac events Grade 3 - 4 | 0
  drug-related infection Grade 3 - 4 | 0
  drug-related sepsis Grade 3 - 4 | 0
  drug-related interstitial lung disease Grade 3 - 4 | 0
  drug-related renal failure Grade 3 - 4 | 2
  drug-related thromboembolic events Grade 3 - 4 | 5
  drug-related febrile neutropenia Grade 3 - 4 | 4

ADVERSE EVENTS:
Time Frame: Day 1 up to 30 days after last dose of study drug. Participants were in the study until disease progression or toxicity/decision by patient-investigator.
Groups:
- Cetuximab + Cisplatin/Vinorelbine: Intravenous (IV) cetuximab, 400mg per meter squared (m²), week 1, then 250mg/m² weekly, until progressive disease (PD) or toxicity or participant-principal investigator (PPI)decision stopped the treatment. One hour of observation required after each infusion. IV cisplatin, 25 mg/m², Day 1 and 8 of each 21 day cycle, Maximum 6 cycles. Pre-cisplatin hydration could begin during 1-hour post cetuximab observation period. IV vinorelbine, 80mg/m², Day 1 of each 21 day cycle, maximum 6 cycles. One cycle was defined as a 21-day treatment period, unless chemotherapy administration was delayed (cycle duration was longer). All study drugs discontinued if participants experienced PD. If unacceptable toxicities to any study drug occurred, any drug could be modified (reduced, delayed, omitted, or discontinued) independently of the other drugs If no PD, cetuximab could be given as monotherapy after completion of the 6 treatment cycles or after early discontinuation of cis/vin due to intolerance.
Arm/Group | Cetuximab + Cisplatin/Vinorelbine
Serious Adverse Events (participants affected / at risk) | 38/60
Other Adverse Events (participants affected / at risk) | 59/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab + Cisplatin/Vinorelbine (N=60)
Clostridium difficile colitis (Infections and infestations) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neutrophil count decreased (Investigations) | 1
Pericardial effusion (Cardiac disorders) | 1
Peritonitis (Infections and infestations) | 1
Renal failure acute (Renal and urinary disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Administration site abscess (Infections and infestations) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Deep vein thrombosis (Vascular disorders) | 3
Diverticular perforation (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Neutropenic infection (Infections and infestations) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Fatigue (General disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8
Disease progression (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Lobar pneumonia (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Renal failure (Renal and urinary disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 1
Tooth infection (Infections and infestations) | 1
Asthenia (General disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mucosal inflammation (General disorders) | 2
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Pneumonia (Infections and infestations) | 1
Atrial fibrillation (Cardiac disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lung infection pseudomonal (Infections and infestations) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab + Cisplatin/Vinorelbine (N=60)
Dry mouth (Gastrointestinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Headache (Nervous system disorders) | 14
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6
Insomnia (Psychiatric disorders) | 19
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 5
Vomiting (Gastrointestinal disorders) | 22
Weight decreased (Investigations) | 15
Alopecia (Skin and subcutaneous tissue disorders) | 9
Constipation (Gastrointestinal disorders) | 31
Cough (Respiratory, thoracic and mediastinal disorders) | 23
Diarrhoea (Gastrointestinal disorders) | 16
Erythema (Skin and subcutaneous tissue disorders) | 6
Hypersensitivity (Immune system disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 16
Localised infection (Infections and infestations) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10
Neuropathy peripheral (Nervous system disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 16
Syncope (Nervous system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Urinary tract infection (Infections and infestations) | 4
Abdominal pain (Gastrointestinal disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 9
Fatigue (General disorders) | 37
Vision blurred (Eye disorders) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4
Depressed mood (Psychiatric disorders) | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 25
Dry eye (Eye disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 12
Hot flush (Vascular disorders) | 5
Hypertrichosis (Skin and subcutaneous tissue disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 7
Nausea (Gastrointestinal disorders) | 41
Non-cardiac chest pain (General disorders) | 3
Pain (General disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 14
Dysgeusia (Nervous system disorders) | 10
Nail disorder (Skin and subcutaneous tissue disorders) | 6
Nail infection (Infections and infestations) | 3
Neutrophil count (Investigations) | 3
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Rhinitis (Infections and infestations) | 3
Asthenia (General disorders) | 9
Blood creatinine increased (Investigations) | 3
Chills (General disorders) | 6
Decreased appetite (Metabolism and nutrition disorders) | 20
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 27
Hypotension (Vascular disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 7
Mucosal inflammation (General disorders) | 12
Peripheral sensory neuropathy (Nervous system disorders) | 11
Pharyngitis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 4
Pyrexia (General disorders) | 11
Tachycardia (Cardiac disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 13
Chest pain (General disorders) | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Infection (Infections and infestations) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 20
Paronychia (Infections and infestations) | 4
White blood cell count decreased (Investigations) | 4
Anxiety (Psychiatric disorders) | 13
Depression (Psychiatric disorders) | 3
Dysuria (Renal and urinary disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Stomatitis (Gastrointestinal disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.